CLINICAL TRIAL: NCT01664936
Title: Non-Invasive Cerenkov Luminescence Imaging of Lymphoma, Leukemia and Metastatic Lymph Nodes
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12-050
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Head and Neck Cancers
Keywords: 18F-FDG PET/CT scan; 131I therapy; Cerenkov Luminescence Imaging; 12-050; Lymphoma; Leukemia; Metastatic Lymph Nodes
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pts receiving a PET/CT scan with Metastatic LNs: This study seeks to optically image the Cerenkov emissions from the PET tracer 18F-FDG and the radiotherapeutic 131I in a cohort of patients with primary tumor sites and from pathologic lymph nodes after routine 18F-FDG PET 31I radiotherapy and/or investigational study scans. We will include a subset of patients with normal lymph nodes during screening. This subset of patients will be imaged as a negative control for this study.
  Interventions: Radiation: Cerenkov emissions from the PET tracer 18F-FDG and the radiotherapeutic 131I

INTERVENTIONS:
Radiation: Cerenkov emissions from the PET tracer 18F-FDG and the radiotherapeutic 131I — We will image (i) patients who are receiving a PET/CT scan for tumors in the head / neck region and (ii) patients with thyroid cancer after 131I radioablation. Two scans will be completed per patient, one of the primary tumors, as well as a 'background' scan of the contralateral side or, if tumor is there as well, of the forearm. The device to be used is an intensified charge-coupled device camera (Stanford Photonics, Palo Alto, CA) connected to a laptop PC. The camera will use a Quartz high-UV transmission 50 mm 0.8f lens. The Imaging device will be placed approximately 5 cm from the area of the patient to be imaged.

SUMMARY:
The purpose of this study is to see if a new way of imaging called the Cerenkov luminescence or effect that is used with a standard clinical PET/CT and/or investigation scans can be done in order to capture tumor sizes. The investigators believe endoscopies and surgical procedures could benefit from this type of imaging in the future. The Cerenkov imaging could be used as a guide for surgical resections.

The purpose of this study is to use the Cerenkov light from FDG, Iodine-131 tracer sand/or other investigational tracers to image tumors and its sizes in the head, neck, breast, axillary and pelvic regions with a highly sensitive camera. The investigators will be trying to see if we can get another picture of the tumor using the Cerenkov light as part of the standard clinical scan or therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age or older.
* Participant is scheduled for standard clinical and/or investigational PET/CT scan or 131I therapy within the Nuclear Medicine Service at Main Hospital.
* Patients must have had pathologic lymph node metastases in the neck, axillary or inguinal area (do not need to be biopsy proven) from either leukemias, lymphomas: , Head and Neck cancers (e.g. tonsillar, nasopharynx, tongue carcinoma, breast cancer or melanoma;or lymphoma or tonsillar or squamous cell carcinoma with metastases in the neck region for PET/CT imaging, or thyroid cancer for thyroid ablation therapy. Any other more infrequent cancer metastasizing with nodal metastasis in the neck, axilla and inguinal regions to cervical lymph nodes is eligible as well as the primary goal is to image pathological (i.e. hypermetabolic) lymph nodes.
* Patients with hypermetabolic activity and uptake in the neck,axilla, breast and inguinal region on scan, defined visually as significant lesion suspicious for malignancy by a nuclear medicine physician or trainee. (We will include a subset of patients with normal lymph nodes during screening. This subset of patients will be imaged as a negative control for this study.)

Exclusion Criteria:

* Patients imaged for Cerenkov luminescence are going to be required to be in a darkened enclosure for at least 10 minutes and sit still during image acquisition, potentially covered by a dark cloth in case that the ambient light level remains too high for the ultra-sensitive camera. Any conditions that would prevent this will exclude the patients.
* There are any other past medical, physiological or demographic concerns. This includes any patients with skin blemishes that are present at the dermis over the tumor, as these are of particular interest for use of this technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC Clinics
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
feasibility of clinical Cerenkov imaging | 2 years
  is to assess the feasibility of clinical Cerenkov luminescence imaging using current clinical radiotracers (18F-FDG and 131I) and a highly sensitive camera.

SECONDARY OUTCOMES:
Correlate Cerenkov imaging | 2 years
  signal with uptake of the radiotracer. Cerenkov images will be correlated with images obtained from standard clinical PET/CT and scintigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Grimm, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/